CLINICAL TRIAL: NCT01386736
Title: Vitamin D Concentrations and Their Effect on Glucose Metabolism in Pediatrics
Brief Title: Vitamin D and Glucose Metabolism in Pediatrics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Maria Vogiatzi, MD, Weill Cornell Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0902010250
Record Dates: First submitted 2011-04-18; First posted 2011-07-01 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Insulin Resistance; Obesity; Vitamin D25 Insufficiency
Keywords: insulin resistance; obesity; adolescence; vitamin D supplementation
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Active Comparator): Subjects will randomly be assigned to Vitamin D drops versus placebo drops.
  Interventions: Drug: Vitamin D drops
- Placebo (Placebo Comparator): Subjects will randomly be assigned to Vitamin D drops versus placebo drops.
  Interventions: Drug: Placebo drops

INTERVENTIONS:
Drug: Vitamin D drops — Subjects will be randomly assigned to Vitamin D 3,000 Units per day or Placebo drops.
  Arms: Vitamin D
Drug: Placebo drops — Subjects will be randomly assigned to Vitamin D 3,000 Units per day or Placebo drops.
  Arms: Placebo

SUMMARY:
The discovery that the vitamin D receptor is expressed in more than 30 tissues indicates that the physiologic functions of vitamin D are much broader than its well-known role in the regulation of calcium absorption and bone metabolism. There is evidence that vitamin D is involved in the pathogenesis of cancer, cardiovascular disease, multiple sclerosis, and type I diabetes. Recent epidemiological evidence points to a strong association between vitamin D insufficiency and insulin resistance, the metabolic syndrome, and type II diabetes. The investigators would like to examine the role of vitamin D in the development of insulin resistance in overweight children and adolescents, which represent a high risk population for cardiovascular and metabolic complications. The investigators propose a prospective randomized clinical trial of vitamin D supplementation in overweight, insulin resistant, vitamin D deficient children. The investigators objective is to assess if changes in insulin resistance, fasting lipid profiles, blood pressure, and inflammatory markers occur in these patients post treatment with vitamin D. Additionally, concomitant changes in calcium and bone metabolism after vitamin D treatment will be evaluated. This is because, contrary to adults, the optimal vitamin D concentrations that regulate calcium and bone metabolism have not been established in pediatrics.

ELIGIBILITY:
Inclusion Criteria:

1. BMI>85th% for age & sex
2. Vitamin D25 between 10-20ng/ml
3. Normal serum Ca concentrations >8.5mg/dl
4. Evidence of insulin resistance (measured by HOMA-IR, and QUICKI indices)

Exclusion Criteria:

1. Vitamin D25<10ng/ml
2. No parental consent
3. No evidence of insulin resistance
4. BMI < 85th percentile
5. Known diagnosis of type 1 or 2 diabetes
6. Severe underlying disease such as liver disease, end-stage renal disease, or malignancy
7. Present medication that affects insulin sensitivity such as steroids or Metformin
8. Any chronic illness or administration of medications that is associated with fat malabsorption as they may interfere with vitamin D absorption.
9. Known history of hypocalcemia, calcium disorder (such as Di George syndrome)
10. Serum Calcium concentration < 8.5mg/dl
11. Other drugs that might effect vitamin D metabolism due to induction of P450 enzyme activity.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
To determine changes in insulin sensitivity induced by vitamin D supplementation in obese children with insulin resistance. | 4 months
  To our knowledge, there are no prospective randomized clinical trials on examining the effects of vitamin D treatment on insulin resistance and bone metabolism in vitamin D deficient, insulin resistant, obese children. We would like to determine if giving Vitamin D supplementation to obese children will help reduce their insulin resistance. We plan to measure Vitamin D levels and HOMA-IR at baseline and compare this to levels post-supplementation. Our timeframe is baseline and 4 months.

SECONDARY OUTCOMES:
To quantify the associations between vitamin D 25 concentration, insulin resistance, and calcium metabolism in overweight children. | 4 months
  The normal values for vitamin D are not standardized. In children, it is generally accepted, that vitamin D25 levels>20ng/ml are indicative of vitamin D sufficiency. Data in adults, however, suggest that this cutoff for vitamin D sufficiency should be raised to greater than 30ng/ml. Analysis of bone metabolism in this study will give some insight to the effects of vitamin D treatment in this population of children, and may help further define acceptable vitamin D levels in determining vitamin D deficiency and insufficiency. Our timeframe is baseline and 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Vogiatzi, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Alemzadeh R, Kichler J, Babar G, Calhoun M. Hypovitaminosis D in obese children and adolescents: relationship with adiposity, insulin sensitivity, ethnicity, and season. Metabolism. 2008 Feb;57(2):183-91. doi: 10.1016/j.metabol.2007.08.023. PMID 18191047
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Chiu KC, Chu A, Go VL, Saad MF. Hypovitaminosis D is associated with insulin resistance and beta cell dysfunction. Am J Clin Nutr. 2004 May;79(5):820-5. doi: 10.1093/ajcn/79.5.820. PMID 15113720
- [Background] Smotkin-Tangorra M, Purushothaman R, Gupta A, Nejati G, Anhalt H, Ten S. Prevalence of vitamin D insufficiency in obese children and adolescents. J Pediatr Endocrinol Metab. 2007 Jul;20(7):817-23. doi: 10.1515/jpem.2007.20.7.817. PMID 17849744
- [Background] Munns C, Zacharin MR, Rodda CP, Batch JA, Morley R, Cranswick NE, Craig ME, Cutfield WS, Hofman PL, Taylor BJ, Grover SR, Pasco JA, Burgner D, Cowell CT; Paediatric Endocrine Group; Paediatric Bone Australasia. Prevention and treatment of infant and childhood vitamin D deficiency in Australia and New Zealand: a consensus statement. Med J Aust. 2006 Sep 4;185(5):268-72. doi: 10.5694/j.1326-5377.2006.tb00558.x. PMID 16948623
- [Background] Keskin M, Kurtoglu S, Kendirci M, Atabek ME, Yazici C. Homeostasis model assessment is more reliable than the fasting glucose/insulin ratio and quantitative insulin sensitivity check index for assessing insulin resistance among obese children and adolescents. Pediatrics. 2005 Apr;115(4):e500-3. doi: 10.1542/peds.2004-1921. Epub 2005 Mar 1. PMID 15741351
- [Background] Katz A, Nambi SS, Mather K, Baron AD, Follmann DA, Sullivan G, Quon MJ. Quantitative insulin sensitivity check index: a simple, accurate method for assessing insulin sensitivity in humans. J Clin Endocrinol Metab. 2000 Jul;85(7):2402-10. doi: 10.1210/jcem.85.7.6661. PMID 10902785
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Background] Radikova Z, Koska J, Huckova M, Ksinantova L, Imrich R, Vigas M, Trnovec T, Langer P, Sebokova E, Klimes I. Insulin sensitivity indices: a proposal of cut-off points for simple identification of insulin-resistant subjects. Exp Clin Endocrinol Diabetes. 2006 May;114(5):249-56. doi: 10.1055/s-2006-924233. PMID 16804799
- [Background] Pittas AG, Lau J, Hu FB, Dawson-Hughes B. The role of vitamin D and calcium in type 2 diabetes. A systematic review and meta-analysis. J Clin Endocrinol Metab. 2007 Jun;92(6):2017-29. doi: 10.1210/jc.2007-0298. Epub 2007 Mar 27. PMID 17389701
- [Background] Palomer X, Gonzalez-Clemente JM, Blanco-Vaca F, Mauricio D. Role of vitamin D in the pathogenesis of type 2 diabetes mellitus. Diabetes Obes Metab. 2008 Mar;10(3):185-97. doi: 10.1111/j.1463-1326.2007.00710.x. PMID 18269634
- [Background] Forouhi NG, Luan J, Cooper A, Boucher BJ, Wareham NJ. Baseline serum 25-hydroxy vitamin d is predictive of future glycemic status and insulin resistance: the Medical Research Council Ely Prospective Study 1990-2000. Diabetes. 2008 Oct;57(10):2619-25. doi: 10.2337/db08-0593. Epub 2008 Jun 30. PMID 18591391